CLINICAL TRIAL: NCT03590782
Title: Erector Spinae Plane Block for Acute Pain Management in Emergency Department Patients With Rib Fractures
Brief Title: Erector Spinae Plane Block for Acute Pain Management in the Emergency Department
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: Dr. Ian Surdhar (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pending
Record Dates: First submitted 2018-07-04; First posted 2018-07-18 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Rib Fractures; Nerve Block
MeSH Terms: conditions — Rib Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Erector Spinae Block — An ultrasound guided erector spinae block will be performed.

SUMMARY:
Rib fractures are a common cause of respiratory distress in trauma patients as poor pain control and subsequent hypoventilation commonly results in lung tissue collapse (atelectasis). The current mainstay of treatment in rib fractures are oral and intravenous opioids however these are often ineffective and can also precipitate hypoventilation. Recently there has been interest in regional anaesthesia techniques for managing painful conditions of the thorax as a way to avoid pain and opioid related hypoventilation. These techniques include ultrasound guided nerve blocks such as the intercostal, paravertebral and serratus anterior blocks. The use of these techniques is however limited by minimal dermatomal coverage as well as a high incidence of complications The erector spinae plane block is a new, very promising technique which offers a safe means of providing anaesthesia to a large part of the hemithorax with a single injection. The proposed study will seek to establish whether the erector spinae plane block can be successfully used in the emergency department for pain control in patients with acute rib fractures.

DETAILED DESCRIPTION:
Rib fractures represent a significant cause of morbidity and mortality in trauma patients. Hypoventilation secondary to pain and altered breathing mechanics frequently leads to respiratory distress and may necessitate admission to an ICU. Currently, opioids are the mainstay of treatment in rib fracture pain management however they are often ineffective and themselves can also promote hypoventilation. A more effective means of analgesia in rib fractures is the use of regional anaesthesia techniques including ultrasound (US) guided nerve blocks. Multiple studies have shown promising results with the use of US guided intercostal nerve blocks, paravertebral blocks and serratus anterior blocks for acute and long-term pain control in rib fractures, however each of these techniques has significant drawbacks including being limited to single dermatomes, high incidence of complications, and incomplete analgesia of the hemithorax. Recently, the erector spinae plane block (ESPB) has come to the forefront as a potential safe and effective option for analgesia in painful conditions of the thorax. This technique involves identifying the erector spinae muscles at the level of a given thoracic transverse process and injecting local anaesthetic into the fascial plane (Figures 1, 2, and 3); the local anaesthetic then spreads through the fascial plane both cephalad and caudad to the injection point and will anaesthetize the thoracic sensory nerves that run in this plane at multiple dermatomal levels (Figure 4). Moreover, because the target point of injection is both superficial and protected by the bony transverse process the incidence of complications is felt to be low. While this technique has been successfully used in the field of anaesthesiology, the ESPB has yet to be integrated into the practice of emergency medicine physicians. In fact, only one paper has detailed it's use for acute pain control in the emergency department (ED; 7). Given the high morbidity associated with rib fractures, the inadequacy of opioid analgesia and the strong safety profile of the ESPB, the proposed study seeks to address whether this block can be used to provide analgesia in ED patients with acute rib fractures. This first study will provide proof of concept that this technique is a useful and safe technique for emergency providers to use.

Objectives To address whether the ESPB can successfully be used for analgesia in ED patients with rib fractures.

Hypothesis The investigators hypothesize that the ESPB will be a safe and effective means of analgesia in ED patients with rib fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* Acute rib fractures with pain that is subjectively poorly controlled despite oral and/or intravenous opioids.

Exclusion Criteria:

* Hemodynamic instability,
* Active infection overlying the site of injection
* Patients receiving anticoagulation
* Patients with a history of a bleeding disorder
* Patients with thrombocytopenia
* Pregnant, are incarcerated
* Decline the procedure
* Inability to provide consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with acute rib fractures failing traditional therapy.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue pain scale | 30-60 minutes
  Pain scale with be taken pre- and post-block and regular intervals. The visual analogue pain scale ranges from 0-10, with 0 being no pain and 10 being the worse pain imaginable. Lower numerical scores are better for outcomes as it implies that the pain is more well managed.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada